CLINICAL TRIAL: NCT02835677
Title: Integrating Caregiver Support Into MS Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Memphis VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2205-P; RX002205 (Other: Memphis VA Medical Center)
Record Dates: First submitted 2016-07-12; First posted 2016-07-18 (Estimated); Results first posted 2019-07-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-05

CONDITIONS: Multiple Sclerosis
Keywords: Caregivers; Activities of Daily Living
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Behavioral intervention with caregivers to reduce stress and management of patient concerns, particularly ambulation
  Interventions: Behavioral: Behavioral

INTERVENTIONS:
Behavioral: Behavioral — Education and skills building, including problem solving, cognitive restructuring, and stress management

SUMMARY:
With loss of mobility in multiple sclerosis (MS) comes an increase in amount and types of caregiver assistance, with a concomitant increase in burden for the caregiver. In fact, effect on caregiver burden can be seen as a potential indicator of the efficacy of MS management, suggesting that the caregiver is an appropriate and independent target for MS therapeutic strategies.

MS patients report difficulty implementing and continuing with home exercise, mobility, and walking programs. This feasibility study will test integration of a successful behavioral caregiving intervention into clinical practice to improve functioning of Veterans with multiple sclerosis (MS) and their Caregivers. Caregivers of Veterans with MS will receive a behavioral caregiver intervention designed to address caregiver coping and management of patient concerns, with special focus on patient mobility and walking. A pre-post intervention design will compare outcomes for Veterans and Caregivers.

For Veterans, the intervention will target Caregiver participation in home-based Veteran mobility activities. MS Caregivers report high burden, stress, and depression involved in caring for their loved ones, especially as mobility declines and these outcomes are related to physical and emotional health status of the patient. For Caregivers, the intervention will focus on improving Caregiver coping and on managing MS-related problems. Outcomes for both will be measured at baseline, 3 months, and 6 months.

Study Objectives include:

* Test whether a caregiver intervention can be integrated into an MS clinical setting.
* Determine whether Caregiver outcomes are improved (depression, burden, anxiety, and number of Veteran MS problems and safety alerts reported).
* Determine whether Veteran outcomes are improved (Expanded Disability Status Scale, timed up and go test, self-efficacy, and depression).
* Determine which types of Caregivers will benefit most.
* Determine which types of Veterans will benefit most.
* Refine materials for future clinical research, translation and implementation.

ELIGIBILITY:
Inclusion Criteria:

* Veteran being seen in MS clinic at Memphis VA
* Veteran ambulatory
* Caregiver/care partner who agrees to participate

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-09-07 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Olivia Nichols, PhD, Principal Investigator — Memphis VA Medical Center, Memphis, TN
Locations (1):
- Memphis VA Medical Center, Memphis, TN, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred in the Neurology Service at the Memphis Veterans Affairs Medical Center (VAMC).
Period: Overall Study
Arm/Group | Intervention
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] — Caregiver
  years | 54.8 (13.3)
Age, Continuous [Mean (Standard Deviation); unit: years] — Care Recipient
  years | 55.9 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Caregiver
  Participants
    Female | 21
    Male | 4
Sex: Female, Male [Count of Participants; unit: Participants] — Care Recipient
  Participants
    Female | 6
    Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Caregiver
  Participants
    Hispanic or Latino | 0
    Not Hispanic or Latino | 25
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25
Marital status [Count of Participants; unit: Participants] — Caregiver
  Participants
    Married | 19
    Not married | 6
Relationship to care recipient [Count of Participants; unit: Participants]
  Spouse | 17
  Parent | 3
  Sibling | 3
  Child | 2
Anxiety change from baseline to six months [Mean (Standard Deviation); unit: units on a scale] — Caregiver, General Anxiety Disorders Scale-7, (GAD-7), range 0-21, lower better Population: Lost to followup
  units on a scale
    Baseline | 5.2 (5.3)
    Six months: number analyzed (Participants) | 23
    Six months | 4.6 (4.4)
Depression change from baseline to six months [Mean (Standard Deviation); unit: units on a scale] — Caregiver, Patient Health Questionnaire - 9, PHQ-9, range 0-27, lower better Population: Lost to followup
  units on a scale
    Baseline | 5.4 (5.2)
    Six months: number analyzed (Participants) | 23
    Six months | 3.7 (4.7)
Burden change from baseline to six months [Mean (Standard Deviation); unit: units on a scale] — Caregiver, Zarit Burden Inventory, 12 item, 0-48, lower better Population: Lost to followup
  units on a scale
    Baseline | 6.6 (6.9)
    Six months: number analyzed (Participants) | 23
    Six months | 7.5 (6.2)
Caregiving tasks change from baseline to six months [Mean (Standard Deviation); unit: units on a scale] — Caregiving Tasks in Multiple Sclerosis Scale (CTiMSS), range 0-96, lower better Population: Lost to followup
  units on a scale
    Baseline | 30.7 (19.9)
    Six months: number analyzed (Participants) | 23
    Six months | 31.0 (19.2)
Social support change from baseline to six months [Mean (Standard Deviation); unit: units on a scale] — Caregiver, received support, satisfaction, negative interactions, range 0-30, higher better Population: Lost to followup
  units on a scale
    Baseline | 18.0 (6.6)
    Six months: number analyzed (Participants) | 23
    Six months | 18.9 (5.3)
Self Care change from baseline to six months [Mean (Standard Deviation); unit: units on a scale] — Caregiver, health services use, range 0-14, higher is better Population: Lost to followup
  units on a scale
    Baseline | 9.4 (2.0)
    Six months: number analyzed (Participants) | 23
    Six months | 10.5 (1.9)
Caregiving frustrations change from baseline to six months [Mean (Standard Deviation); unit: units on a scale] — Feel like yelling or hitting, range 0-4, lower better Population: Lost to followup
  units on a scale
    Baseline | 0.7 (0.7)
    Six months: number analyzed (Participants) | 23
    Six months | 0.6 (0.7)
Hours on duty change from baseline to six months [Mean (Standard Deviation); unit: hours] — Mahoney Vigilance Scale, number of hours caregiver feels on duty, range 0-24 Population: Lost to followup
  hours
    Baseline | 12.3 (8.9)
    Six months: number analyzed (Participants) | 23
    Six months | 12.0 (9.8)
Hours performing tasks change from baseline to six months [Mean (Standard Deviation); unit: hours] — Mahoney Vigilance Scale, number of hours actually performing tasks, range 0-24 Population: Missing data, Lost to followup
  hours
    Baseline: number analyzed (Participants) | 24
    Baseline | 3.4 (2.5)
    Six months: number analyzed (Participants) | 23
    Six months | 4.3 (3.7)
Concerning care recipient behaviors change from baseline to six months [Mean (Standard Deviation); unit: number of behaviors reported] — Number of possible patient troubling behaviors or concerns, range, 0-27 Population: Lost to followup
  number of behaviors reported
    Baseline | 9.5 (4.7)
    Six months: number analyzed (Participants) | 23
    Six months | 8.0 (5.3)
Number of behaviors that bother change from baseline to six months [Mean (Standard Deviation); unit: number of behaviors] — Number of possible patient troubling behaviors or concerns that bother the caregiver, range 0-27 Population: Lost to followup
  number of behaviors
    Baseline | 6.1 (5.5)
    Six months: number analyzed (Participants) | 23
    Six months | 3.9 (4.1)
Timed Up and Go Test change from baseline to six months [Mean (Standard Deviation); unit: seconds] — Care Recipient, Timed Up and Go Test (TUGT), seconds (for analysis - square root transformed seconds), fewer better Population: Missing data
  seconds
    Baseline: number analyzed (Participants) | 23
    Baseline | 4.2 (1.6)
    Six months: number analyzed (Participants) | 19
    Six months | 4.1 (2.2)
MS Self-efficacy change from baseline to six months [Mean (Standard Deviation); unit: units on a scale] — Care Recipient, Multiple Sclerosis Self-Efficacy Scale (MSSS), score 14-84, higher better Population: Missing data
  units on a scale
    Baseline: number analyzed (Participants) | 23
    Baseline | 52.3 (10.8)
    Six months: number analyzed (Participants) | 24
    Six months | 54.0 (12.6)
Disability Scale change from baseline to six months [Count of Participants; unit: Participants] — Care Recipient, Expanded Disability Status Scale (EDSS),0-10, lower better. Categories are percentage with mild (0-2.5 points), moderate (3.0-5.0), and severe (> 6) disability. Population: Missing data
  Participants
    Baseline: number analyzed (Participants) | 24
    Baseline: Mild | 12
    Baseline: Moderate | 4
    Baseline: Severe | 8
    Six monts: number analyzed (Participants) | 23
    Six monts: Mild | 11
    Six monts: Moderate | 3
    Six monts: Severe | 9
Depression change from baseline to six months [Mean (Standard Deviation); unit: units on a scale] — Care Recipient, Patient Health Questionnaire - 9, PHQ-9, range 0-27, lower better Population: Missing data
  units on a scale
    Baselinw | 7.5 (5.5)
    Six months: number analyzed (Participants) | 24
    Six months | 7.9 (5.8)
Employment, full or part time [Count of Participants; unit: Participants] — Caregiver
  Participants | 11
Employment, full or part time [Count of Participants; unit: Participants] — Care Recipient
  Participants | 12

OUTCOME MEASURES:

1. Primary Outcome: Depression Measured With the Patient Health Questionnaire 9 (PHQ-9) Scale
Description: Caregiver primary outcome. PHQ-9, range 0-27, lower better
Time Frame: baseline, 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 25
units on a scale
  Baseline | 5.2 (1.1)
  Six month | 4.6 (0.9)

2. Primary Outcome: Burden Measured With the Zarit Burden Inventory
Description: Caregiver primary outcome. Zarit Burden Inventory, 12 item, 0-48, lower better
Time Frame: baseline, 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 25
units on a scale
  Baseline | 6.6 (1.4)
  Six month | 7.5 (1.3)

3. Primary Outcome: Anxiety Measured With the Generalized Anxiety Disorders 7 Scale
Description: Caregiver primary outcome. General Anxiety Disorders Scale - GAD-7, range 0-21, lower better
Time Frame: baseline, 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 25
units on a scale
  Baseline | 5.2 (1.1)
  Six month | 4.6 (0.9)

4. Primary Outcome: Number of Patient MS Problems
Description: Caregiver primary outcome - number of possible troubling patient problems and concerns, range 0-27, lower better
Time Frame: baseline, 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 25
units on a scale
  Baseline | 9.5 (0.9)
  Six month | 7.9 (1.1)

5. Primary Outcome: Bother With Patient MS Problems
Description: Number of troubling patient problems or concerns that bother the caregiver, range 0-27, lower better
Time Frame: Baseline, 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 25
units on a scale
  Baseline | 6.1 (1.1)
  Six months | 3.9 (0.8)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-01): https://cdn.clinicaltrials.gov/large-docs/77/NCT02835677/Prot_SAP_000.pdf